CLINICAL TRIAL: NCT01676831
Title: A Phase I/IIa, Dose-Ranging Safety and Efficacy Study of Topical Resiquimod for the Treatment of Early Stage Cutaneous T Cell Lymphoma
Brief Title: Topical Resiquimod for the Treatment of Early Stage Cutaneous T Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 813320(UPCC03411); 1R01FD004092-01A1 (FDA); NCT01497795 (obsolete NCT alias)
Record Dates: First submitted 2012-07-15; First posted 2012-08-31 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- topical resiquimod 0.06% (Experimental): Topical resiquimod 0.06% will be applied in dosing frequencies that are periodically adjusted to tolerability. Dosing frequency will be 3 times a week. The dosing frequency may be adjusted (1,2,3,5,or 7times per week) based on the physician assessment of tolerability. Treatment will occur for 8 weeks followed by 4 weeks rest followed by another 8 weeks of treatment with 4 weeks rest. At 24 weeks a final evaluation will be performed. Those with a partial response at week 24 will have the option to continue therapy for up to another 12 weeks.
  Interventions: Drug: Topical resiquimod 0.06%
- topical resiquimod 0.03% (Experimental): Topical resiquimod 0.03% will be applied in dosing frequencies that are periodically adjusted to tolerability. Dosing frequency will begin 5 times a week. The dosing frequency may be adjusted (1,2,3,5,or 7times per week) based on the physician assessment of tolerability. Treatment will occur for 8 weeks followed by 4 weeks rest followed by another 8 weeks of treatment with 4 weeks rest. At 24 weeks a final evaluation will be performed. Those with a partial response at week 24 will have the option to continue therapy for up to another 12 weeks.
  Interventions: Drug: topical resiquimod 0.03%

INTERVENTIONS:
Drug: Topical resiquimod 0.06% — topical resiquimod 0.06% dosing frequency begins at 3 times per week and evaluated every two weeks. Will be applied for a total of 8 weeks followed by 4 weeks rest and then followed by another 8 weeks of application with another 4 weeks rest.
  Arms: topical resiquimod 0.06%
Drug: topical resiquimod 0.03% — topical resiquimod 0.03% applied initially 5 times weekly for 8 weeks with adjustments up or down based upon tolerability followed by 4 weeks rest followed by another 8 weeks of treatment followed by another 4 week rest period.
  Arms: topical resiquimod 0.03%

SUMMARY:
The objective of this study is to explore the safety and the preliminary efficacy of two concentrations (0.06% and 0.03%)gel that is applied to lesions of early stage (IA, IB,IIA) Cutaneous T Cell Lymphoma patients.

This study is supported by grant 1R01FD004092-01A1 from the Office of Orphan Products Development, FDA.

DETAILED DESCRIPTION:
This is an open-label, dose-ranging study in subjects with early stage (IA, IB, 2A) CTCL. Patients with early stage CTCL will be screened for eligibility. Eligible subjects will be enrolled in up to 2 treatment groups of up to 8 subjects each.

Treatment groups will be:

1. Resiquimod 0.06% will be applied in dosing frequencies that are periodically adjusted according to tolerability. Subjects will begin dosing at 3 times per week (3x/wk), and will be evaluated at the clinic every two weeks. The dosing frequency (1, 2, 3, 5, or 7x/wk) may be adjusted in a stepwise manner after each two week interval based on the physician assessment of tolerability (maintained, increased, decreased with or without a dosing interruption [rest period]). Resiquimod will be applied for 8 weeks (COT1) followed by a 4 week no-treatment period. If the subject has not required permanent discontinuation from treatment, the subject will repeat a second course of treatment of 8 weeks (COT2) followed by a 4 week no-treatment period. Subjects will apply up to 500 mg of study drug per day based upon the total surface area that is treated (~250 mg of product / 50 cm2 of lesion surface area).
2. Resiquimod 0.03% applied as described for Treatment Group 1. However, initial applications will be 5 times per week with the dosing frequency adjusted upward as tolerated every two weeks.

The initial cohort will be assigned to Treatment Group 1. After 4 subjects have completed at least 4 weeks of dosing, a safety review meeting will be conducted by a committee consisting of the P.I., a biostatistician, and at least one other physician familiar with CTCL responses. The Safety Review Committee (SRC) will determine, based on the review of the tolerability data, the starting concentration/frequency of the next group of 4 subjects.

For a given subject the concentration assignment (0.06% or 0.03%) will remain the same (only frequency may vary). It is planned that approximately 8 subjects will be enrolled in each group.

A treatment regimen will be considered inadequately tolerated if 2 or more subjects within the treatment cohort require protocol mandated permanent discontinuation. Treatment regimens for newly enrolled subjects and/or of current subjects on treatment will be adjusted accordingly per protocol. The Safety Review Committee (SRC) will determine the occurrence of any dose-limiting toxicities (DLTs), defined below in Section 6.4.6. A subsequent phase II study will further explore efficacy of the MTD in an expanded study.

Up to 2 subjects per Treatment Group who discontinue from the study due to reasons unrelated to safety reasons (e.g. personal, lost to follow-up, etc) may be replaced.

The investigator will determine the target CTCL lesions and treatment area. During each COT, subjects will treat at least 1 but no more than 4 target lesions in the 0.06% dosing group and no ,more than 5 target lesions in the 0.03% treatment group with a total combined treatment area that is ≥25 cm2 but ≤100 cm2. Unless a lesion is considered to have completely resolved by clinical assessment at 4 weeks post COT1 (PCOT1), subjects will treat the same baseline target lesions throughout the COT1 and COT2. The amount of drug applied per dose during each COT may vary depending on the total size of the target lesions but may not exceed 500 mg per day.

For COT1, subjects will be evaluated at baseline, Week 2, 4, 6, 8 and 12 (PCOT1). For COT2, subjects will be evaluated at Week 12 (PCOT1/COT2 baseline) 14, 16, 18, 20 and 24 (4 weeks post COT2, PCOT2). The End of study (EOS) will be at PCOT2, or if a subject permanently discontinues study drug prematurely, at 4 weeks after the last dose.

Rest periods from treatment may be instituted by the investigator as needed to manage tolerance, with resumption of treatment upon adequate resolution per investigator discretion.

Subjects in both treatment groups who experience a partial response but not a complete response at week 24 can continue treatment for up to another 12 weeks with the same concentration.

During this time they will be evaluated every 4 weeks up to 12 weeks. At that time they will have a 4 week rest period and then a final evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Males or female ≥18 years of age at the time of study enrollment
2. Have a clinical diagnosis of cutaneous T cell lymphoma CTCL, including documentation of a skin biopsy with histological findings consistent with CTCL (atypical epidermotrophic or folliculocentric T-cells). Unconfirmed diagnosis of CTCL must have a biopsy to confirm at screening
3. Have Stage IA, IB or IIA: T1 or T2 (patches or plaques) with measurable lesions.
4. Previous treatment with at least one standard therapy used to treat Stage IA, IB or IIA CTCL including but not limited to oral corticosteroids, high-potency topical corticosteroids, topical mechlorethamine, topical bexarotene, PUVA, UVB, total body electron beam radiation, biological response or oral methotrexate.
5. Have measurable skin disease with at least 1 to 4 eligible baseline target lesions with a total area >25 cm2 but <100 cm2. Eligible lesions must be below the neck and may not involve the genitalia, intertriginous areas, internally, or to frankly ulcerated or infected skin.
6. Generally healthy other than for CTCL, or with other stable diseases/conditions that are adequately controlled.
7. Willing and able to provide written informed consent.
8. Willing and able to adhere to the protocol requirements, including but not limited to study drug dosing, study drug visits, medication and treatment restrictions, and laboratory tests.
9. Willing and able to discontinue concomitant medications or treatments for CTCL during the study.
10. If a female of child bearing potential, willing to use adequate contraception (defined as double-method contraception, e.g. oral contraceptive usage by subject and condom by partner). Non-child bearing potential is defined as being at least 2 years post-menopausal or being surgically sterile.
11. Willing to abstain from therapeutic sunbathing, tanning beds, etc. for the duration of the study.

Exclusion Criteria:

1. Have a known allergy to resiquimod or any of the excipients in the study drug.
2. Stage IIB or greater CTCL.
3. Require immediate treatment for progressive CTCL.
4. Are unable to discontinue current treatment for CTCL due to risk of progression.
5. Within 8 weeks of treatment initiation (Day 0), have received treatment with:

   * Total body electron beam radiation
   * Investigational drugs or treatments
6. Within 4 weeks of treatment initiation (Day 0), have received treatment with:

   * Local radiation therapy
   * UVB therapy
   * PUVA
   * Any topical chemotherapy
   * Photopheresis
   * Systemic retinoids, corticosteroids, immune response modifiers including imiquimod, interferon inducers, chemotherapeutic agents, biologic agents including interferon
   * Topical corticosteroids or retinoids
7. Within 2 weeks of treatment initiation (Day 0), have received at or adjacent to the target treatment lesions.

   * Any surgical procedures other than biopsies related to CTCL diagnosis or follow-up
   * Any topical treatment other than bland moisturizers (creams, lotions, emollients, etc).
8. Have other concurrent cutaneous conditions in the treatment area or immediately adjacent to the treatment area that would be exacerbated by resiquimod or interfere with assessments.
9. Have a grade 2 or greater laboratory abnormalities (CTCAE v4) at baseline for any of the following:

   * Hemoglobin
   * White blood cell count
   * Platelet count
   * Alanine transferase
   * Aspartate transferase
   * Creatinine
10. Have a known history of or a positive serologic test for infection with human immunodeficiency virus or human T lymphotrophic virus.
11. Are pregnant or nursing, or intending to become pregnant within the duration of the study.
12. Have any clinically significant medical conditions that are unstable, progressive, or inadequately controlled in the opinion of the investigator, that would pose a potential risk for the subject, result in poor compliance with the study requirements, or require treatment with an excluded medication or treatment during the study.
13. Have an active chemical or alcohol dependency as assessed by the investigator.
14. Have systemic collagen vascular disorder, systemic autoimmune disease, an organ transplant or diagnosis of cancer within 5 years other than CTCL (not including basal cell carcinoma, non-invasive squamous cell cancer of the skin, malignant melanoma in situ, or cervical carcinoma in situ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2015-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain H Rook, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rook AH, Gelfand JM, Wysocka M, Troxel AB, Benoit B, Surber C, Elenitsas R, Buchanan MA, Leahy DS, Watanabe R, Kirsch IR, Kim EJ, Clark RA. Topical resiquimod can induce disease regression and enhance T-cell effector functions in cutaneous T-cell lymphoma. Blood. 2015 Sep 17;126(12):1452-61. doi: 10.1182/blood-2015-02-630335. Epub 2015 Jul 30. PMID 26228486

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topical Resiquimod 0.06% | Topical Resiquimod 0.03%
Started | 8 | 5
Completed | 8 | 4
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Resiquimod 0.06% | Topical Resiquimod 0.03% | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants That Tolerated the Maximum Drug Dose
Description: After four subjects have completed at least four weeks of study drug dosing a safety review meeting will be conducted by a safety review committee. No subjects will be enrolled in the next concentration (0.03%)group until all eight have been evaluated in the 0.06% group.
  The safety review committee reviews all patient data including adverse events to indicate whether the patient can escalate to the highest dose.
Time Frame: after 4 subjects have completed 4 weeks of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Resiquimod 0.06% | Topical Resiquimod 0.03%
Number analyzed (Participants) | 8 | 4
Participants | 8 | 4

2. Secondary Outcome: Secondary End Points: Efficacy- CAILDS SCORE
Description: The secondary endpoint is:
  • The Response Rate (Complete or Partial Response) based on Composite Assessment of Index Lesions Disease Severity (CAILDS) score at EOS for the baseline target lesions. Complete Response is defined as a score of '0' on the CAILDS scale. Partial response is defined as a reduction of at least 50% in the CAILDS. The outcome measure will indicate how many received complete response (CR), partial response (PR), and stable disease (SD).
Time Frame: Up to 24 weeks or At the conclusion of patient therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Resiquimod 0.06% | Topical Resiquimod 0.03%
Number analyzed (Participants) | 8 | 4
Participants
  Complete Response (CR) | 4 | 0
  Partial Response (PR) | 3 | 2
  Stable Disease (SD) | 1 | 2

3. Secondary Outcome: Secondary End Points: Efficacy- SWAT SCORE
Description: The secondary endpoint is:
  The total surface area of involvement will also be assessed (SWAT score). A partial response will represent improvement in 50% or greater of the skin surface area with regression of lesions. A complete response will represent complete clear clearing of skin lesions and in the case of stage IIA patients, resolution of lymphadenopathy. The outcome measure will indicate how many received complete response (CR), partial response (PR), and stable disease (SD).
Time Frame: Up to 24 weeks or At the conclusion of patient therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Resiquimod 0.06% | Topical Resiquimod 0.03%
Number analyzed (Participants) | 8 | 4
Participants
  Complete Response (CR) | 2 | 0
  Partial Response (PR) | 5 | 2
  Stable Disease (SD) | 1 | 2

ADVERSE EVENTS:
Time Frame: through study completion (3years)
Description: Patient was assessed at each study visit.
Groups:
- Topical Resiquimod 0.03%: Topical resiquimod 0.03% will be applied in dosing frequencies that are periodically adjusted to tolerability. Dosing frequency will begin 5 times a week. The dosing frequency may be adjusted (1,2,3,5,or 7times per week) based on the physician assessment of tolerability. Treatment will occur for 8 weeks followed by 4 weeks rest followed by another 8 weeks of treatment with 4 weeks rest. At 24 weeks a final evaluation will be performed. Those with a partial response at week 24 will have the option to continue therapy for up to another 12 weeks.
  topical resiquimod 0.03%: topical resiquimod 0.03% applied initially 5 times weekly for 8 weeks with adjustments up or down based upon tolerability followed by 4 weeks rest followed by another 8 weeks of treatment followed by another 4 week rest period.
  13 patients were consented and enrolled. 1 patient dropped out of the clinical study this patient was in the 0.03% arm of the study. As such 5 patients were measured for adverse events
Arm/Group | Topical Resiquimod 0.06% | Topical Resiquimod 0.03%
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 6/8 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Resiquimod 0.06% (N=8) | Topical Resiquimod 0.03% (N=5)
fever (Immune system disorders) | 2 (2) | 0 (0)
skin erosion (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
headache (General disorders) | 2 (2) | 0 (0)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
myalgia (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes